CLINICAL TRIAL: NCT06000384
Title: Investigate if Ultrasound is Comparable to Chest X-ray in Verification of Intensive Care Patients Enteral Feeding Tube Positioning in an Observational Study
Brief Title: Is Ultrasound Comparable to Chest X-ray in Verification of Intensive Care Patients Enteral Feeding Tube Positioning.
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 590270
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Patient
Keywords: Intensive care patient; Enteral feeding tube

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate methodological if ultrasound is comparable to chest X-ray in verification of intensive care patients enteral feeding tube positioning.

The main question to answer is: Is ultrasound a comparable method to chest X-ray in verification of intensive care patients enteral feeding tube positioning.

DETAILED DESCRIPTION:
In Norway, around 4000 patients are yearly in need of ventilator, and many of them will need enteral nutrition through a feeding tube. 40 % of all intensive care patients have signs of malnutrition. If ultrasound is a comparable method to chest X-ray in verification of intensive care patients enteral feeding tube positioning, then enteral nutrition in many cases can be started several hours earlier than using chest X-ray verification. The ultrasound examination will be performed in a research based in a 4-step approach. In this project 20-30 intensive care patients prescribed by a medical physician to have an enteral feeding tube will be included in the project due to written informed consent by 1) Awake intensive care patient or by 2) Patients informal caregiver if the patient is not competent to consent.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patient prescribed by a medical physician to have an enteral feeding tube

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients in need of enteral tube feeding
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Measuring enteral tube position both by standard chest X-ray and ultrasound | maximum five minutes for each method
  Ultrasound measure by a research based 4-step approach

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lie, Professor, Principal Investigator — Norwegian University of Science and Technology - NTNU.
Locations (1):
- Lillehammer sykehus, Sykehuset Innlandet, Lillehammer, Innlandet, Norway